CLINICAL TRIAL: NCT05857891
Title: The Effect of Erythropoietin on Alveolar Fluid Clearance in Patients With Acute Respiratory Distress Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2018-11-134
Record Dates: First submitted 2023-04-24; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Erythropoietin; ARDS; Lung Water Clearance
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erythropoietin group (Experimental): intravenous injection of 40000iu of rhEPO
  Interventions: Drug: Human erythropoietin injection
- 0.9%NS (Placebo Comparator): intravenous injection of the same volume of 0.9%NS as the test group
  Interventions: Drug: 0.9%NaCl

INTERVENTIONS:
Drug: Human erythropoietin injection — Each subject in the test group received 40000iu of human erythropoietin intravenously
  Other Names: Treatment measures taken according to the patient's condition
  Arms: Erythropoietin group
Drug: 0.9%NaCl — Each subject in the control group was injected with an equal volume of 0.9%NaCl
  Other Names: Treatment measures taken according to the patient's condition
  Arms: 0.9%NS

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a common acute and critical disease in clinic. The clinical mortality is as high as 30%-40%. At present, there is no specific treatment. Erythropoietin (EPO), also known as erythrocyte- stimulating factor, erythropoietin, has a certain amount in normal human body, mainly synthesized by liver in infants and kidneys in adults, which can stimulate erythropoiesis. In recent years, more and more studies have shown that high-dose exogenous EPO administration has benefit effects on multi-organ protection. Therefore, we designed this prospective, double-blind, placebo-controlled trial for defecting EPO on the alveolar fluid clearance of ARDS. The study mainly answers the following questions: Does human erythropoietin accelerate the resolution of alveolar edema in ARDS? Is there any effect on hospital survival? The study will draw conclusions by comparing the control group with the experimental group.

DETAILED DESCRIPTION:
This study was designed as a double-blind, randomized controlled trial. Neither the subject nor the investigator knew the allocation of treatment drugs. Subjects signed the informed consent form, completed all screening assessments, and were randomized in the order of screening eligibility after screening eligibility. The investigator or designee generated the corresponding case number and drug number using a simple randomization method. Information about the subject's trial product allocation was placed in an emergency envelope and retained by the investigator for use in an emergency. Randomised subjects who withdraw from the clinical trial for any reason, regardless of whether they have taken the trial medication, will retain their case number and medication number and will not be allowed to re-enter the trial.

The investigator participating in this trial is a clinician with appropriate experience, who can make treatment decision based on the clinical response and laboratory test results of the subject. The specific process of the study is as follows:

1. The subjects of this study were patients with ARDS admitted to ICU.
2. After signing the informed consent form, complete medical history collection, vital signs and detailed physical examination will be performed. Patients meeting the inclusion criteria but not meeting the exclusion criteria will be randomized into the study.
3. Patients with ARDS who met the inclusion criteria were connected to PiCCO, randomly assigned to the following two groups, and monitored continuously for 3 days. Group A: Erythropoietin, 40000 IU, single intravenous injection. Group B: 0.9%NaCl group, with the same volume as group A, single intravenous injection.
4. The baseline values of extravascular lung water index (EVLWI) and pulmonary vascular permeability index (PVPI) were monitored by PiCCO after recording the general conditions of the subjects included in the study before intervention. After EPO or 0.9% NaCl intervention, EVLWI and PVPI at 0, 6, 12, 24, 48 and 72h after EPO or normal saline administration, and blood gas analysis, CRP, PCT, blood routine, inflammatory factors (TNF-a,IL-6,IL-8,IL-1β), endothelial cell injury marker (s-ICAM-1), alveolar epithelial cell injury marker (sRAGE,SP-D) and other laboratory indicators and clinical indicators such as peak airway pressure, mean airway pressure and positive end-expiratory pressure (PEEP) at 0, 1, 2 and 3 days after administration were recorded. The hospital survival rate and 28-day survival rate were compared between the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years;
* Meeting diagnostic criteria for sepsis 3.0;
* Tracheal intubation and mechanical ventilation;
* Meeting the diagnostic criteria of ARDS Berlin;
* Willing to accept treatment and sign an informed consent form;

Exclusion Criteria:

* Age <18 years;
* Pregnancy or lactation;
* Patients with malignant tumors;
* Recombinant human erythropoietin (rhEPO) allergic patients;
* Hemoglobin (Hb) ≥120g/L;
* have recently taken rhEPO (within 3 months) or participated in other clinical trials;
* History of thromboembolic disease (pulmonary embolism, heart attack, cerebral infarction, arteriovenous thrombosis);
* Inability or unwillingness to provide informed consent or to comply with the requirements of the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
EVLWI | Changes of EVLWI at 0,6,12,24 ,48 and 72 hours after intervention
  extravascular lung water index
PVPI | Changes of PVPI at 0,6,12,24 ,48 and 72 hours after intervention
  pulmonary vascular permeability index

SECONDARY OUTCOMES:
Survival rate | 28-day hospital survival
  28-day survival rate
Oxygenation index | Changes of oxygenation index at 0, 1, 2 and 3 days after intervention
  PaO2/FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Ye Gao, PhD, Study Director — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- SAHWenzhouMU, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Wiese L, Hempel C, Penkowa M, Kirkby N, Kurtzhals JA. Recombinant human erythropoietin increases survival and reduces neuronal apoptosis in a murine model of cerebral malaria. Malar J. 2008 Jan 7;7:3. doi: 10.1186/1475-2875-7-3. PMID 18179698
- [Result] Gantner DC, Bailey M, Presneill J, French CJ, Nichol A, Little L, Bellomo R; EPO-TBI Investigators; the ANZICS Clinical Trials Group. Erythropoietin to Reduce Mortality in Traumatic Brain Injury: A Post-hoc Dose-effect Analysis. Ann Surg. 2018 Mar;267(3):585-589. doi: 10.1097/SLA.0000000000002142. PMID 28151802
- [Result] Tsai TH, Lu CH, Wallace CG, Chang WN, Chen SF, Huang CR, Tsai NW, Lan MY, Sung PH, Liu CF, Yip HK. Erythropoietin improves long-term neurological outcome in acute ischemic stroke patients: a randomized, prospective, placebo-controlled clinical trial. Crit Care. 2015 Feb 25;19(1):49. doi: 10.1186/s13054-015-0761-8. PMID 25888250
- [Result] Yip HK, Tsai TH, Lin HS, Chen SF, Sun CK, Leu S, Yuen CM, Tan TY, Lan MY, Liou CW, Lu CH, Chang WN. Effect of erythropoietin on level of circulating endothelial progenitor cells and outcome in patients after acute ischemic stroke. Crit Care. 2011;15(1):R40. doi: 10.1186/cc10002. Epub 2011 Jan 26. PMID 21269484
- [Result] Ozawa T, Toba K, Suzuki H, Kato K, Iso Y, Akutsu Y, Kobayashi Y, Takeyama Y, Kobayashi N, Yoshimura N, Akazawa K, Aizawa Y; EPO/AMI-I Pilot Study Researchers. Single-dose intravenous administration of recombinant human erythropoietin is a promising treatment for patients with acute myocardial infarction - randomized controlled pilot trial of EPO/AMI-1 study -. Circ J. 2010 Jul;74(7):1415-23. doi: 10.1253/circj.cj-10-0109. Epub 2010 May 22. PMID 20501957
- [Result] Voors AA, Belonje AM, Zijlstra F, Hillege HL, Anker SD, Slart RH, Tio RA, van 't Hof A, Jukema JW, Peels HO, Henriques JP, Ten Berg JM, Vos J, van Gilst WH, van Veldhuisen DJ; HEBE III Investigators. A single dose of erythropoietin in ST-elevation myocardial infarction. Eur Heart J. 2010 Nov;31(21):2593-600. doi: 10.1093/eurheartj/ehq304. Epub 2010 Aug 29. PMID 20802250
- [Result] Tsai TH, Lu CH, Wallace CG, Chang WN, Chen SF, Huang CR, Tsai NW, Lan MY, Sung PH, Liu CF, Yip HK. Erratum to: Erythropoietin improves long-term neurological outcome in acute ischemic stroke patients: a randomized, prospective, placebo-controlled clinical trial. Crit Care. 2016 Mar 31;20:78. doi: 10.1186/s13054-016-1256-y. No abstract available. PMID 27037155
- [Result] Suhs KW, Hein K, Sattler MB, Gorlitz A, Ciupka C, Scholz K, Kasmann-Kellner B, Papanagiotou P, Schaffler N, Restemeyer C, Bittersohl D, Hassenstein A, Seitz B, Reith W, Fassbender K, Hilgers R, Heesen C, Bahr M, Diem R. A randomized, double-blind, phase 2 study of erythropoietin in optic neuritis. Ann Neurol. 2012 Aug;72(2):199-210. doi: 10.1002/ana.23573. PMID 22926853
- [Result] Corwin HL, Gettinger A, Fabian TC, May A, Pearl RG, Heard S, An R, Bowers PJ, Burton P, Klausner MA, Corwin MJ; EPO Critical Care Trials Group. Efficacy and safety of epoetin alfa in critically ill patients. N Engl J Med. 2007 Sep 6;357(10):965-76. doi: 10.1056/NEJMoa071533. PMID 17804841
- [Result] Kakavas S, Demestiha T, Vasileiou P, Xanthos T. Erythropoetin as a novel agent with pleiotropic effects against acute lung injury. Eur J Clin Pharmacol. 2011 Jan;67(1):1-9. doi: 10.1007/s00228-010-0938-7. Epub 2010 Nov 11. PMID 21069520
- [Result] Rocha J, Eduardo-Figueira M, Barateiro A, Fernandes A, Brites D, Pinto R, Freitas M, Fernandes E, Mota-Filipe H, Sepodes B. Erythropoietin reduces acute lung injury and multiple organ failure/dysfunction associated to a scald-burn inflammatory injury in the rat. Inflammation. 2015 Feb;38(1):312-26. doi: 10.1007/s10753-014-0035-7. PMID 25270658
- [Result] Tascilar O, Cakmak GK, Tekin IO, Emre AU, Ucan BH, Bahadir B, Acikgoz S, Irkorucu O, Karakaya K, Balbaloglu H, Kertis G, Ankarali H, Comert M. Protective effects of erythropoietin against acute lung injury in a rat model of acute necrotizing pancreatitis. World J Gastroenterol. 2007 Dec 14;13(46):6172-82. doi: 10.3748/wjg.v13.i46.6172. PMID 18069756
- [Result] MacRedmond R, Singhera GK, Dorscheid DR. Erythropoietin inhibits respiratory epithelial cell apoptosis in a model of acute lung injury. Eur Respir J. 2009 Jun;33(6):1403-14. doi: 10.1183/09031936.00084608. Epub 2009 Jan 22. PMID 19164355
- [Result] Heeschen C, Aicher A, Lehmann R, Fichtlscherer S, Vasa M, Urbich C, Mildner-Rihm C, Martin H, Zeiher AM, Dimmeler S. Erythropoietin is a potent physiologic stimulus for endothelial progenitor cell mobilization. Blood. 2003 Aug 15;102(4):1340-6. doi: 10.1182/blood-2003-01-0223. Epub 2003 Apr 17. PMID 12702503
- [Result] Shang Y, Li X, Prasad PV, Xu S, Yao S, Liu D, Yuan S, Feng D. Erythropoietin attenuates lung injury in lipopolysaccharide treated rats. J Surg Res. 2009 Jul;155(1):104-10. doi: 10.1016/j.jss.2008.10.003. Epub 2008 Nov 8. PMID 19285686
- [Result] Ware LB, Matthay MA. Alveolar fluid clearance is impaired in the majority of patients with acute lung injury and the acute respiratory distress syndrome. Am J Respir Crit Care Med. 2001 May;163(6):1376-83. doi: 10.1164/ajrccm.163.6.2004035. PMID 11371404
- [Result] Phillips CR, Chesnutt MS, Smith SM. Extravascular lung water in sepsis-associated acute respiratory distress syndrome: indexing with predicted body weight improves correlation with severity of illness and survival. Crit Care Med. 2008 Jan;36(1):69-73. doi: 10.1097/01.CCM.0000295314.01232.BE. PMID 18090369